CLINICAL TRIAL: NCT05552417
Title: Efficacy of Pectointercostal Facial Nerve Block for Postoperative Pain Management After Sternotomy in Pediatric Open Cardiac Surgery:A Randomized Controlled Trial
Brief Title: Pectointercostal Block for Postoperative Pain Management After Sternotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Elhaddad, Lecturer of Anesthesia, ICU and Pain managment, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-92-2022
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Conventional control group(C) (n=--) where --- children will not receive any intervention.
- Pectointercostal (Active Comparator): Pectointercostal facial group (PI) (n=--) where --children will have bilateral Pectointercostal Block.
  Interventions: Other: Pectointercostal facial plan block

INTERVENTIONS:
Other: Pectointercostal facial plan block — Pectointercostal facial group (PI) (n=--) where --children will have bilateral Pectointercostal Block.
  Other Names: Pectointercostal facial nerve block
  Arms: Pectointercostal

SUMMARY:
This randomized, controlled study is designed to assess the quality of analgesia provided by ultrasound-guided bilateral pectointercostal facial block in children undergoing cardiac surgery via midline sternotomy.

DETAILED DESCRIPTION:
Following approval from the research and ethics committee ,preoprrative preparation, and induction of anesthesia The patient will be assigned to two equal groups. Conventional control group(C) (n=30) where --- children will not receive any intervention.

Pectointercostal facial group (PI) (n=30) where --children will have bilateral Pectointercostal Block.

Patient positioning and preparation for Ultrasound-guided PIFB After skin disinfection, the PIFB will be performed in a supine position using a high-frequency (6-13 MHz) linear ultrasound probe (S-NerveTM; SonoSite Inc., Bothell, WA, USA). The probe will be placed at 2 cm lateral from the sternum and parallel to the sternum and will be scanned laterally to identify 4th and 5th costal cartilage The pecto-intercostal fascial plane will be located between the pectoralis major muscle and the external intercostal muscle or the costal cartilage. A 22G, 50 mm peripheral block needle, Stimuplex® Ultra 360 (B. Braun, Melsungen, Germany) will be placed under the pectoralis major and above the external intercostal muscle with an in-plane approach with the ultrasound probe, in a caudal-to-cranial direction until the tip is positioned in the interfascial plane between the PMM and IIM .

A test bolus of saline (1 mL) will be injected to determine that the tip has been placed in the correct fascial layers. Finally, 1.5 mg/kg of 0.2% bupivacaine will be injected into this plane in two locations, over the 2nd and 4th rib. The method on the other side of the PIFB will be the same Care will be taken not to cross the toxic dose of bupivacaine (3 mg/kg). (6) .

Heart rate, mean arterial pressure, and oxygen saturation will be monitored continuously.

After completion of the surgery, inhalational anesthetics will be stopped as well as the muscle relaxant.

The patient will be then transferred to the ICU.Postoperative assessment and analgesic regimen: An IV Paracetamol 15 mg / kg will be given and will be repeated every 8 hours .The Face, Legs, Activity, Cry, Consolability scale (FLACC) (table 1) will be assessed in the PICU and every 4 hours for 24 hours. The time to the first request of rescue postoperative analgesic will be: "the time interval between the onset of block and the first request to postoperative analgesia". When patients first complain of pain (FLACC score ≥4) rescue analgesia will be given in the form of incremental intravenous morphine

ELIGIBILITY:
Inclusion Criteria:

* age 6 to 36 months
* sex both
* Weight > 5kg
* Pathology A-V canal , ASD closure, VSD closure surgery through a midline sternotomy.

Exclusion Criteria:

* Redo patient.
* History of allergic reactions to local anesthetics.
* Bleeding disorders with INR > 1.5 and/or platelets < 50 000.
* Rash or signs of infection at the injection site.
* Emergency procedures.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Post-operative pain score | At 4 hours.
  Post-operative pain score by The Face, Legs, Activity, Cry, Consolability scale ( Each category is scored on a 0-2 scale, which results in a total score of 0-10 0:comfortable,1-3:Mild discomfort,4-6:Moderate discomfort, &7-10:Sever discomfort ) (FLACC) scale pain score at 4 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided